CLINICAL TRIAL: NCT07285616
Title: Optimizing Graft Selection in Glaucoma Surgery
Brief Title: Optimizing Graft Selection in Glaucoma Surgery: A Comparative Study of Sclera, Pericardium, and Corneal Tissue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00157655
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma
Keywords: PRESERFLO; surgery; MicroShunt
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- PreserFlo with Donor Scleral Patch Graft (Experimental): Participants undergo PreserFlo MicroShunt implantation with a donor scleral patch graft covering the tube. Standard perioperative care (e.g., MMC/5-FU per site protocol) and scheduled follow-up (day 1; week 1-2; months 1, 3, 6, 9, 12). Outcomes include IOP, hypotony, tube erosion, conjunctival complications, infection, reoperations, device longevity, patient-reported comfort/cosmesis, and resource use. Primary and revision cases are included per stratified randomization.
  Interventions: Procedure: MicroShunt with Scleral Patch Graft
- PreserFlo with Corneal Patch Graft (Experimental): Participants undergo PreserFlo MicroShunt implantation with a donor corneal patch graft covering the tube. Standard perioperative care and identical follow-up schedule. Outcomes as above: IOP control, complications (including erosion and hypotony), reoperations, longevity, patient-reported outcomes, and resource use. Primary and revision cases are included per stratified randomization.
  Interventions: Procedure: MicroShunt with Corneal Patch Graft
- PreserFlo with Pericardial Patch Graft (Experimental): Participants undergo PreserFlo MicroShunt implantation with a pericardial patch graft covering the tube. Standard perioperative care and identical follow-up schedule. Outcomes as above: IOP control, complication profile, reoperations, longevity, patient-reported outcomes, and resource use. Primary and revision cases are included per stratified randomization.
  Interventions: Procedure: MicroShunt with Pericardial Patch Graft

INTERVENTIONS:
Procedure: MicroShunt with Scleral Patch Graft — Placement of PreserFlo MicroShunt with donor scleral patch graft to cover the tube.
  Arms: PreserFlo with Donor Scleral Patch Graft
Procedure: MicroShunt with Corneal Patch Graft — Placement of PreserFlo MicroShunt with donor corneal patch graft to cover the tube.
  Arms: PreserFlo with Corneal Patch Graft
Procedure: MicroShunt with Pericardial Patch Graft — Placement of PreserFlo MicroShunt with pericardial patch graft to cover the tube.
  Arms: PreserFlo with Pericardial Patch Graft

SUMMARY:
Glaucoma refers to a group of progressive optic neuropathies that lead to permanent vision loss. Glaucoma is the leading cause of irreversible blindness globally. In 2020, it was estimated to affect 76 million individuals worldwide, with projections indicating this number will rise to 111.8 million by 2040. In Canada, glaucoma affects an estimated 2.7-7.5% of individuals over the age of 50, contributing substantially to the national disease burden. This condition is linked to damage of the optic nerve due to elevated intraocular pressure (IOP; raised eye pressure), which results in the loss of retinal ganglion cells. Therefore, most of the treatments are guided towards reducing the IOP either via using laser, medications or surgery.

Glaucoma surgery is typically reserved for cases where IOP remains uncontrolled while on maximum tolerated medical therapy and/or where glaucoma progression warrants surgery. The goal of many glaucoma surgeries is to divert aqueous humor from the anterior chamber to the subconjunctival space, therefore reducing intraocular pressure. The device used for this purpose are the PRESERFLO™ MicroShunt (Glaukos Corporation, Laguna Hills, CA, USA) (the documents will interchangeably use terms "stent" and "shunt" to refer to these devices in the text below). The device is implanted using the ab externo approach to channel fluid from the anterior chamber to the subconjunctival/subtenon space. To reduce postoperative fibrosis and inhibit fibroblast activity that could obstruct flow and lead to device failure, 5-fluorouracil (5-FU) or mitomycin C (MMC) are administered. Additionally, a double-layered closure of conjunctiva and Tenon's is performed to minimize Tenon's migration and blockage of tenon the stents. Despite these measures, stent encapsulation and failure are still too common requiring revisions and bleb needling in 2-20% of cases within the first 12 months of follow-up.

This project will involve a series of studies evaluating graft selection in PreserFlo MicroShunt implantation, focusing on donor sclera, cornea, and pericardium as patch graft materials. First, the investigators will conduct a prospective, randomized study comparing clinical outcomes between these graft types. Outcomes of interest will include surgical success rates, post-operative hypotony, tube erosion, conjunctival complications, infection, and overall device longevity. Donor sclera has long been used as a patch graft in glaucoma drainage device surgery and is associated with low erosion rates and reliable long-term results. Corneal tissue is increasingly used due to its transparency and availability through eye banks, with demonstrated safety in ocular surface reconstruction and tube coverage. Pericardium is another durable, biocompatible option, historically applied in both cardiovascular and ocular surgery, and has shown effectiveness as a patch graft in glaucoma drainage implants. This comparison will extend to both primary implantation and revision surgeries, recognizing the high clinical relevance of graft performance in complex cases.

Building on these results, the investigators will then perform a cost-effectiveness analysis of graft strategies, incorporating surgical time, post-operative management, complication rates, and need for re-operation. An economic model will be developed to evaluate costs and resource utilization associated with each material, providing valuable data for policy and surgical decision-making. Finally, the investigators will conduct a patient-reported outcome (PRO) study to assess patient comfort and satisfaction with different grafts. Surveys will evaluate domains such as foreign body sensation, cosmesis, and overall satisfaction at key time points (immediate post-operative period, 1 week, 3 weeks, and 3 months). These results will highlight the patient perspective, an often underrepresented but critical factor in surgical innovation.

Together, these studies will comprehensively assess graft selection from surgical, economic, and patient-centered perspectives, informing evidence-based practice in glaucoma care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Patients selected for PreserFlo microshunt surgery and XEN stent alone or in combination with cataract surgery.
3. Ability to comprehend the study procedures

Exclusion Criteria:

1. Unwilling or unable to give consent
2. Unable to come for scheduled post-operative visits
3. Pregnant or nursing women
4. Previous cyclodestructive procedures, scleral buckling procedures, or presence of silicone oil
5. Conjunctival scarring precluding a glaucoma surgery superiorly
6. Active iris neovascularization or active proliferative retinopathy
7. Vitreous in the anterior chamber for which a vitrectomy is anticipated.
8. Previous trabeculectomy, tube-shunt implantation, or surgeries that shunt aqueous outflow into the subconjunctival space

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Intraocular Pressure (IOP) from Baseline to 12 Months | 12 months
  IOP measured by Goldmann applanation tonometry (mmHg) at baseline, post-operative Day 1, Week 1, Month 1, Month 3, Month 6, and Month 12. The primary endpoint will be the mean change at 12 months.
Surgical Success Rate at 12 Months | 12 months
  Proportion of eyes achieving target IOP (≤18 mmHg or ≥20% reduction from baseline) without additional glaucoma surgery, vision-threatening complication, or device removal.

SECONDARY OUTCOMES:
Glaucoma medication burden | 12 months
  Number of glaucoma medications used per patient, counted from the medication list at each follow-up (baseline, Month 3, 6, 12). Outcome reported as: Mean change in number of medications.
Need for re-operation | 12 months
  Number and percentage of eyes requiring any additional glaucoma or device-related surgery during the study period.
  Outcome reported as: Count and proportion of eyes re-operated.
Bleb needling rate | 12 months
  Number and proportion of eyes requiring bleb needling postoperatively to maintain or restore filtration.
Tube/patch graft exposure or erosion | 12 months
  Clinically confirmed exposure or erosion of tube or patch graft, as documented on slit-lamp exam.
  Outcome reported as: Number and percentage of affected eyes.
Hypotony | 12 months
  IOP < 5 mmHg on two consecutive visits measured by Goldmann applanation tonometry (mmHg).
  Outcome reported as: Number and percentage of eyes meeting the definition.
Infection | 12 months
  Any endophthalmitis, blebitis, or wound infection confirmed on clinical exam. Outcome reported as: Number and percentage of eyes with infection.
Best-corrected visual acuity (BCVA) change | 12 months
  BCVA measured using a standard Early Treatment Diabetic Retinopathy Study (ETDRS) chart at 4 m (logMAR scale).
  Outcome reported as: Mean change in logMAR from baseline to 12 months (lower values = better vision).
Device survival (time to failure) | Up to 12 months
  Time from surgery to defined surgical failure (loss of pressure control, device removal, or re-operation).
  Outcome reported as: Kaplan-Meier survival curve; median time to failure.
Patient-reported comfort | Immediate postop (day 1), 1 week, 3 weeks, 3 months.
  Measured using a Visual Analog Scale (VAS, 0-10) where 0 = no discomfort and 10 = worst possible discomfort.
  Assessment points: Post-op Day 1, Week 1, Week 3, and Month 3. Outcome reported as: Mean ± SD at each time point.
Foreign body sensation | Day 1, 1 week, 3 weeks, 3 months.
  Evaluated using a Likert scale (1-5) where 1 = none and 5 = severe sensation. Assessment points: Day 1, Week 1, Week 3, Month 3. Outcome reported as: Mean ± SD and proportion reporting moderate-to-severe sensation (≥4).
Cosmesis/satisfaction | 3 weeks and 3 months.
  Measured with a 5-point Likert scale assessing satisfaction with postoperative appearance (1 = very dissatisfied; 5 = very satisfied).
  Assessment points: Week 3 and Month 3. Outcome reported as: Mean ± SD; higher scores = greater satisfaction.
Health care resource use | 12 months
  Number of postoperative visits, additional procedures, and unscheduled urgent encounters recorded per participant from the medical record.
  Outcome reported as: Mean count per participant and associated cost estimate (CAD).
Cost-utility | 12 months
  Calculated using trial-based costs and quality-adjusted life-year (QALY) estimates derived from EQ-5D-5L utility weights.
  Outcome reported as: Incremental cost per QALY gained by graft type.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No